CLINICAL TRIAL: NCT01616589
Title: Acquisition of Saliva Samples for Validation as a Specimen Type in the Esoterix Genetic Laboratories Fragile X Assay
Brief Title: Validation of Saliva in the Esoterix Genetic Laboratories Fragile X Assay
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Esoterix Genetic Laboratories, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GGFX0001
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X syndrome; Fragile X full mutation; Fragile X premutation; Fragile X intermediate; CGG repeat length
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In some cases, the de-identified, residual saliva specimen may be used in quality assurance; it may be used in clinical testing as a control; it may be used for future research studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fragile X full mutation (affected): Individual whose previous blood specimen was tested at Esoterix Genetic Laboratories and molecular analysis for fragile X revealed >200 CGG repeats with abnormal methylation pattern; interpretation is full mutation for fragile X syndrome
- Fragile X premutation (carriers): Individual whose previous blood specimen was tested at Esoterix Genetic Laboratories and molecular analysis for fragile X revealed 55-200 CGG repeats with normal methylation pattern; interpretation is premutation carrier of fragile X syndrome
- Fragile X intermediate: Individual whose previous blood specimen was tested at Esoterix Genetic Laboratories and fragile X molecular analysis revealed 45-54 CGG repeats; interpretation is intermediate, not a carrier of a fragile X expansion mutation

SUMMARY:
The purpose of this research is to determine if saliva samples can be used as an alternate sample type to test for fragile X. By using saliva instead of blood, it would be easier for patients to have fragile X testing.

DETAILED DESCRIPTION:
Saliva samples will be prospectively collected from subjects who have previously been tested by Esoterix Genetic Laboratories, LLC using blood specimens and diagnosed as fragile X intermediates, premutations (carriers) or full mutations (affected). Results from fragile X testing with saliva will be compared to results from the blood sample that was previously submitted to Esoterix Genetic Laboratories for testing.

Data from this study will be used for regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

* Subject has previously been identified through molecular testing at Esoterix Genetic Laboratories as a Fragile X intermediate, premutation (carrier) or full mutation (affected).
* In the opinion of the subject's physician, the subject is medically stable and able to provide the required quantity of saliva.
* If Subject is at least 18 years of age:
* Subject must be willing to give written informed consent
* Subject must be willing to comply with the collection procedure
* If Subject is under 18 years of age, the legally authorized representative must give written informed consent and agree to comply with study procedures.

Exclusion Criteria:

* Subject has been determined to be an individual with a normal FMR1 gene.
* Subject has a known medical condition that would cause risk to the donor or, if relevant, the fetus as a result of saliva collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fragile X full mutations (affecteds), fragile X premutations (carriers), and fragile X intermediates who previously had fragile X testing through Esoterix Genetic Laboratories. Subject population will be in the US.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Scholl, PhD, Principal Investigator — Esoterix Genetic Laboratories, LLC
Locations (1):
- Integrated Genetics, Westborough, Massachusetts, United States